CLINICAL TRIAL: NCT02356770
Title: Randomized Controlled Clinical Study to Investigate Effectiveness and Safety of a Collagen Matrix 10808 for Soft Tissue Volume Augmentation After Implant Placement in Single Tooth Gaps
Brief Title: A Clinical Study to Investigate Collagen Matrix 10808 for Soft Tissue Volume Augmentation Around Single Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10860; DRKS00003586 (Registry Identifier: Deutsches Register Klinischer Studien); CIV-11-12-003323 (Other: EUDAMED)
Record Dates: First submitted 2014-12-18; First posted 2015-02-05 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Tooth Loss; Soft Tissue Deficiency
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagen Matrix 10808 (Experimental): Mucosal split-thickness flap in combination with the Collagen Matrix 10808.
  Interventions: Device: Collagen Matrix 10808
- Connective tissue graft (gold standard) (Other): Mucosal split-thickness flap in combination with the connective tissue graft.
  Interventions: Procedure: Connective tissue graft

INTERVENTIONS:
Device: Collagen Matrix 10808 — At the day of the Intervention (day 0) sulcular incisions will be made around the neighbouring teeth and a straight incision from the lingual/palatal line angle of the distal tooth to the lingual/palatal line angle of the mesial tooth. A full thickness flap will be elevated on the lingual side, whereas a split flap will be made at the buccal aspect preparing a soft tissue pouch without the preparation of horizontal release incisions. The Collagen Matrix 10808 will then be positioned in the pouch under the elevated buccal flap. A horizontal mattress suture will be made to immobilize graft to the flap followed by four to five single sutures to close the wound.
  Arms: Collagen Matrix 10808
Procedure: Connective tissue graft — At the day of the Intervention (day 0) sulcular incisions will be made around the neighbouring teeth and a straight incision from the lingual/palatal line angle of the distal tooth to the lingual/palatal line angle of the mesial tooth. A full thickness flap will be elevated on the lingual side, whereas a split flap will be made at the buccal aspect preparing a soft tissue pouch without the preparation of horizontal release incisions. The Connective tissue graft (Gold Standard) will then be positioned in the pouch under the elevated buccal flap. A horizontal mattress suture will be made to immobilize graft to the flap followed by four to five single sutures to close the wound.
  Arms: Connective tissue graft (gold standard)

SUMMARY:
The objective of this study is to investigate the safety and the function of the collagen Matrix 10808 in humans and to compare it versus the standard therapy, the transplantation of the autologous connective tissue graft. The Collagen Matrix was developed for soft tissue augmentation. It is a three dimensional porous Matrix and consists mainly of Collagen I and III.

Study patients must have a single tooth gap with insufficient soft tissue volume after implant placement. Therefore a soft tissue augmentation will be necessary.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effectiveness of soft tissue volume augmentation procedures using the autogenous soft tissue graft or the Collagen Matrix 10808 to gain mucosal thickness. Second the safety of the two procedures will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Implant placement at least 6 weeks and maximum 6 months prior enrolment
2. Necessity of soft tissue augmentation in single tooth gap
3. 2 teeth adjacent to each side of the defect have a mean BOP (Bleeding of probing) of < 30%
4. Basic periodontal examination (BPE <2)
5. 18 years or older
6. Ability to comply with the study-related procedures such as exercising good oral hygiene and attending all follow-up procedures
7. Ability to fully understand the nature of the proposed surgery and ability to sign the informed consent form

Exclusion Criteria:

1. Heavy smoker (> 10 cigarettes per day)
2. Probing depth greater than 4 mm
3. Insulin dependent diabetes
4. General contraindications for dental and/or surgical treatment
5. History of malignancy, radiotherapy, or chemotherapy for malignancy within the past five years
6. Women of child bearing age, not using a standard accepted method of birth control
7. Pregnancy or breast feeding
8. Previous and concurrent medication affecting mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs)
9. Disease affecting connective tissue metabolism (e.g. collagenases).
10. Allergy to collagen
11. Participation in a clinical trial within the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Gain in mucosal soft tissue thickness at day 90 compared to day 0 (Baseline) value measured by trans-mucosal probing | at day 90 compared to day 0 (Baseline)

SECONDARY OUTCOMES:
Assessment of Adverse Events | from Day 0 to Day 90
Closure of the wound | at Day 7, 30, 90
Presence of Swelling | at Day 7, 30, 90
Oral health impact profile (OHIP-G14) score | at day 0, 7, 90
Daily Mefenaminacid consumption | between Day 0 and Day 7
Evaluation of pain using a VAS(Visual Analogue Scale) score daily | between Day 0 and day 7 and at Day 30 and 90
Surgery time | at surgery
Qualitative histological assessment regarding matrix degradation and safety parameters | at day 90
Gain in mucosal soft tissue thickness by 3D volumetric analysis | at day 90, compared to day 0
Gain in mucosal soft tissue thickness measured by trans-mucosal probing | at day 30 compared to day 0
Keratinized Tissue width (mm) | at day 0 and at day 90
Probing Depth (mm) | at day 0 and at day 90
Clinical Attachment Level (mm) | at day 0 and at day 90
Bleeding of Probing (0/1) | at day 0 and at day 90
Plaque Index (0-3) | at day 0 and at day 90
Recession depth (mm) | at day 0 and at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Uebersax, PhD, Study Director — Geistlich Pharma AG
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- Available data/document: 1. Publication: PMID: 27310522 — https://www.ncbi.nlm.nih.gov/pubmed/27310522 — A first publication was published concerning the primary outcome of the transmucosal measurements.
- Available data/document: 2. publicaton: PMID: 28107560 — https://www.ncbi.nlm.nih.gov/pubmed/28107560 — 2. publication concerning the volumetric changes of the soft tissue